CLINICAL TRIAL: NCT02140268
Title: A Phase 1, Single-center, Fixed-sequence, Open Label Study to Evaluate the Effect of Oral Repeated Doses of AZD1722 on the Pharmacokinetics of Oral Midazolam in Healthy Volunteers
Brief Title: To Evaluate the Effect of AZD1722 on the Pharmacokinetics of Oral Midazolam in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5613C00003
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers
Keywords: Phase I; Healthy; Pharmacokinetics
MeSH Terms: interventions — Midazolam; tenapanor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Midazolam 7.5 mg (Active Comparator): Volunteers will receive Midazolam 7.5 mg administered by mouth as a syrup
  Interventions: Drug: Midazolam
- AZD1722 15 mg (Experimental): Volunteers will received AZD1722 15 mg administered by mouth, as a tablet
  Interventions: Drug: AZD1722
- AZD1722 15 mg and Midazolam 7.5 mg (Experimental): Volunteers will receive AZD1722 15 mg tablet and Midazolam 7.5 mg syrup, by mouth
  Interventions: Drug: AZD1722 and Midazolam

INTERVENTIONS:
Drug: Midazolam — Volunteers will receive a single dose of Midazolam 7.5 mg on Day 1
  Arms: Midazolam 7.5 mg
Drug: AZD1722 — Volunteers will receive twice daily, oral doses of AZD1722 15 mg on Days 2-14
  Arms: AZD1722 15 mg
Drug: AZD1722 and Midazolam — On Day 15 volunteers will receive AZD1722 15 mg and Midazolam 7.5 mg at the same time in the morning. In the evening on Day 15 AZD1722 15 mg will be administered alone.
  Arms: AZD1722 15 mg and Midazolam 7.5 mg

SUMMARY:
A Study to Evaluate the Effects of oral repeated doses of AZD1722 on the Pharmacokinetics of Oral Midazolam in Healthy Volunteers

DETAILED DESCRIPTION:
A Phase 1, Single-center, Fixed-sequence, Open Label Study to Evaluate the Effect of Oral Repeated Doses of AZD1722 on the Pharmacokinetics of Oral Midazolam in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:Have a body mass index (BMI) ≥18 and ≤30 kg/m2 and weigh at least 50 kg and no more than 100 kg. Females of non-childbearing potential must be postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the postmenopausal range or documentation of irreversible surgical sterilization by hysterectomy, bilateraloophorectomy or bilateral salpingectomy but not tubal ligation

Females of childbearing potential must have a negative pregnancy test at screening, Day -1, and Day 14 and must not be lactating and use effective contraceptive methods to avoid pregnancy during the treatment period

Male healthy volunteers with a partner of childbearing potential must agree to avoid fathering a child, and refrain from donating sperm, from the first day of dosing until at least 3 months after last dose of the investigational product, and therefore be either sterile or agree to use approved methods of contraception

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the principal investigator, may either put the healthy volunteer at risk because of participation in the study, or influence the results or the healthy volunteer's ability to participate in the study. History or presence of GI, hepatic or renal disease including GI surgery other than appendectomy or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs. Loose stools (BSFS of 6 or 7) ≥2 days in the past 7 days before investigational product administration. Use of medications that are known to affect stool consistency and/or GI motility, including fiber supplements, anti-diarrheals, prokinetic drugs, enemas, probiotic medications or supplements, or salt or electrolyte supplements containing sodium, potassium, chloride, or bicarbonate formulations during the past 7 days before the investigational product administration. Use of any prescribed or non-prescribed medication including antacids, analgesics other than paracetamol/acetaminophen, herbal remedies, vitamins and minerals during the 2 weeks prior to the first administration of investigational product or longer if the medication has a long half-life. Use of drugs or substances with enzyme-inducing properties within 4 weeks prior to the first administration of investigational product.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of midazolam when administered after AZD1722 by assessment of area under the concentration-time curve (AUC) and maximal plasma concentration (Cmax) of midazolam | Blood samples are collected predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 15 and 24 hours post dose on Day 1 and Day 15
  Change in plasma area under the concentration-time curve (AUC) and maximal plasma concentration (Cmax) of midazolam after AZD1722 administration

SECONDARY OUTCOMES:
• To evaluate the pharmacokinetics of the metabolites 1-OH-midazolam and 4-OH-midazolam when midazolam is administered after AZD1722 by assessment of AUC and Cmax of 1-OH-midazolam and 4-OH-midazolam | Blood samples are collected predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 15 and 24 hours post dose on Day 1 and Day 15
  Change in plasma area under the concentration-time curve (AUC) maximal plasma concentration (Cmax) of 1-OH-midazolam and 4-OH-midazolam after AZD1722 administration
To evaluate the pharmacodynamic outcomes of AZD1722 by assessment of how AZD1722 effects stool consistency and frequency | Stool frequency and stool consistency will be measured daily (Day -1 through Day 16)
  Pharmacodynamic outcome of the effect on stool consistency and frequency
To evaluate the plasma concentrations of AZD1722 | Blood samples are collected predose, 1, 2, 4 hours post morning dose on Day 15
  plasma concentrations of AZD1722 to be measured (no PK parameters derived)
To evaluate the pharmacokinetics of midazolam metabolites when administered after AZD1722 by assessment of area under the concentration-time curve (AUC) maximal plasma concentration (Cmax) of 1-OH-midazolam and 4-OH-midazolam | Blood samples are collected predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 15 and 24 hours post dose on Day 1 and Day 15
  Change in plasma area under the concentration-time curve (AUC) maximal plasma concentration (Cmax) of 1-OH-midazolam and 4-OH-midazolam after AZD1722 administration

OTHER OUTCOMES:
To evaluate the safety of AZD1722 when administered with midazolam in terms of adverse events, vital signs, electrocardiogram (ECG), hematology, clinical chemistry, urinalysis and physical examination | Safety assessments performed through the screening period (Day -28) to 10 days after the last dose (Day 16)
  Safety assessments in terms of adverse events, vital signs, electrocardiogram (ECG), hematology, clinical chemistry, urinalysis and physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States